CLINICAL TRIAL: NCT03935633
Title: Phase Ib Clinical Study to Assess the Safety, Tolerability and Pharmacokinetic Parameters of CN128 Tablets to Administration in Thalassemia Patients Aged 16 and Above
Brief Title: Short-term Clinical Study of CN128 in Thalassemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zede Pharma-Tech Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D160605-2
Record Dates: First submitted 2019-04-18; First posted 2019-05-02 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2019-12

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Dosage (Experimental): The dose of CN128 is 20 mg/kg bw， bid.
  Interventions: Drug: CN128 Tablets
- Second Dosage (Experimental): The dose of CN128 is 15 mg/kg bw， bid.
  Interventions: Drug: CN128 Tablets

INTERVENTIONS:
Drug: CN128 Tablets — Iron chelator， oral tablets

SUMMARY:
1. Primary objectives:

   * To study the tolerance and safety of multiple oral administration of CN128 in patients with thalassemia aged 16 years and above.
   * To study the pharmacokinetics of CN128 in thalassemia patients aged 16 and above by multiple oral administrations of CN128
2. Design:

   The study is designed as a safety, tolerability and pharmacokinetic parameters study, phase Ib trial.

   The study is consisted of: multiple dose tolerance and safety study; multiple administration pharmacokinetics.
3. Subject inclusion criteria:

   * Thalassemia patients with serum ferritin ≥ 500 µg/L
   * Patients aged 16 and above
   * HB≥80 g/L before administration
   * Voluntarily participate in the experiment, and the process of obtaining informed consent met the requirements of GCP.
4. Subject exclusion criteria:

   * Hepatitis B surface antigen positive, hepatitis B core antibody positive and HBV-DNA positive, hepatitis C anti-HCV positive, HIV positive, Treponema pallidum positive
   * History of active digestive tract diseases (including gastric ulcer, duodenal ulcer, gastroesophageal varices, ulcerative colitis, Crohn's disease, digestive tract tumors, familial genetic polyps), history of digestive tract perforation, history of digestive tract surgery and influence on drug absorption, and other investigators believe that patients with potential intestinal complications
   * Liver dysfunction (ALT or AST > 2.5×ULN); or renal dysfunction (serum creatinine > 1.5×ULN)
   * Uncontrolled active infections
   * Patients currently taking CYP3A strong inducer or inhibitor drugs or drugs that may prolong the QT interval without temporary suspension of use or temporary substitution of the said drugs
   * ect.
5. Usage:

   All subjects fasted prior to administration of study drug using 240 ml warm water. The people can not drink water within 1h before administration.
6. Pharmacokinetic assessment of CN128 administration:

   PK parameters of CN128 include AUC 0-t, AUC 0-∞, Cmax, Tmax, t1/2, CL/F, Vd/ F, MRT, λz, Css-av, Css-min, Css-max, Accumulation rate, Fluctuation index, etc.
7. Safety and tolerability assessments:

   Evaluation was based on the incidence rate of adverse events (AE) after the administration, study termination information, vital signs, physical examination, laboratory tests and ECG.
8. Statistics

DETAILED DESCRIPTION:
1. Primary objectives:

   * To study the tolerance and safety of multiple oral administration of CN128 in patients with thalassemia aged 16 years and above.
   * To study the pharmacokinetics of CN128 in thalassemia patients aged 16 and above by multiple oral administrations of CN128
2. Design:

   The study is designed as a safety, tolerability and pharmacokinetic parameters study, phase Ib trial.

   The study is consisted of:

   • Multiple dose tolerance and safety study: The trial will start with the lower dose of CN128 given to 8 subjects (20 mg/kg body weight [bw], bid).The dose of second group is 15 mg/kg bw, bid (n=8).

   • Multiple administration pharmacokinetics: AUC 0-t, AUC 0-∞, Cmax, Tmax, t1/2, CL/F, Vd/ F, MRT, λz, Css-av, Css-min, Css-max, Accumulation rate, Fluctuation index, etc.
3. Subject inclusion criteria:

   * Thalassemia patients with serum ferritin ≥ 500 µg/L
   * Patients aged 16 and above
   * HB≥80 g/L before administration
   * Voluntarily participate in the experiment, and the process of obtaining informed consent met the requirements of GCP.
4. Subject exclusion criteria:

   * Hepatitis B surface antigen positive, hepatitis B core antibody positive and HBV-DNA positive, hepatitis C anti-HCV positive, HIV positive, Treponema pallidum positive
   * History of active digestive tract diseases (including gastric ulcer, duodenal ulcer, gastroesophageal varices, ulcerative colitis, Crohn's disease, digestive tract tumors, familial genetic polyps), history of digestive tract perforation, history of digestive tract surgery and influence on drug absorption, and other investigators believe that patients with potential intestinal complications
   * Liver dysfunction (ALT or AST > 2.5×ULN); or renal dysfunction (serum creatinine > 1.5×ULN)
   * Uncontrolled active infections
   * Patients currently taking CYP3A strong inducer or inhibitor drugs or drugs that may prolong the QT interval without temporary suspension of use or temporary substitution of the said drugs
   * Allergic constitution: allergic to or with contraindication of main ingredients or excipients of CN128 tablets (microcrystalline cellulose, cross-linked sodium carboxymethyl cellulose, silica, sodium stearate fumarate, Opadry)
   * Patients who have abnormal ECG with clinical significance: congenital long QT syndrome or known family history of long QT syndrome; QTc > 450ms (male) or QTc > 470ms (female); patients who have ventricular or atrial tachyarrhythmia with clinical significance, etc
   * Family planning participants (including male subjects) during or within three months after the trial
   * Patients with a history of blood donation within 3 months before the trial
   * Patients with a history of smoking (more than 5 cigarettes or products with equivalent nicotine per day), alcoholism (more than 14 units of alcohol per week: 1 alcohol unit equals 10 mL or 8 g pure alcohol; 25 mL 40% liquor, 330 mL 5% beer, 175 mL 12% red wine equals 1.0, 1.5, 2.0 alcohol units respectively), drug abuse and addiction history
   * Patients who smoke, drink or eat any food containing alcohol, xanthine or grapefruit (including chocolate, tea, coffee or cola drinks) within 48 h before using of test drug
   * The subjects should not join in other clinical drug or instrument study or some other clinical studies within 3 months before taking the study drug, except for non interventional studies;
   * Patients with positive results of nicotine and urine drug screening
   * Patients with difficulty in venous blood collection
   * Patients with positive blood pregnancy test results
   * Any patient with conditions which the investigators resume inappropriate to participate in this study, such as: poor health status, poor compliance, unwillingness or inability to comply with treatment regimens, including delayed visits
5. Usage:

   Subjects started fasting for solid from 21:00 on the day before the study and for liquid within 1 h before and after the administration. Subjects in each dose group received a single administration on the first day of the study on an empty stomach. Blood samples were collected at different time points before and within 48 hours after the administration (before the administration on day 3). No administration was conducted on day 2. continuous administration was conducted from day 3 to day 8, twice a day, once in the morning on an empty stomach, once in 12 hours (±15min). The valley concentration blood samples were collected in the morning on day 6, 7 and 8. In the morning of day 9, a single administration was conducted on an empty stomach. Blood samples were taken at the different time points before and within 48 hours after the administration on day 9. Each dose was taken with 240 mL warm water.Except for the water taken together with the tablets, it should be ensured that the water was banned for 1 hour before and after the valley concentration blood sample collection from day 6 to day 8 and 1 hour before and after the administration in the morning on day 1 and day 9.
6. Pharmacokinetic assessment of CN128 administration:

   PK parameters of CN128 include AUC 0-t, AUC 0-∞, Cmax, Tmax, t1/2, CL/F, Vd/ F, MRT, λz, Css-av, Css-min, Css-max, Accumulation rate, Fluctuation index, etc.
7. Safety and tolerability assessments:

   Evaluation was based on the incidence rate of adverse events (AE) after the administration, study termination information, vital signs (including body temperature, pulse, breathing, sitting blood pressure) and physical examination (including height, weight, general condition, skin, neck (including thyroid), eyes, ears, nose, throat, chest, abdomen, back, lymph nodes, limbs and nervous system examinations, and laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function, serum iron, thyroid gland and parathyroid gland function), ECG to evaluate the status.
8. Statistics:

   * Pharmacokinetic analysis:

Phoenix WinNonlin software (Pharsight Corporation, version 7.0) was used to estimate and analyze the parameters of PK in non-atrioventricular model according to dosage. The pharmacokinetic parameters were calculated in real time to fully reflect the characteristics of drug absorption, distribution, metabolism and excretion in human body. The PK parameters of each participant were calculated according to the following methods. PK parameters include:

AUC0-t, AUC0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRT, λz, Css_av, Css_min, Css_max, Accumulation rate and Fluctuation index.

Descriptive statistics were summarized on untransformed datas of drug concentration in plasma at each time point: AUC0 t, AUC0-∞, Cmax, Tmax, t1/2, CL/F, Vd/F, MRTλz, Css_av, Css_min, Css_max, R and DF. Descriptive statistics was used in the analysis of Number (N), arithmetic mean, geometric mean, standard deviation (SD), CV, minimum, median and maximum. Average and individual time-concentration curves were drawn according to the study group.

• Safety analysis All AE, treatment emergent adverse events (TEAE), drug-related TEAE, grade 3 or above TEAE, serious adverse events (SAE), drug-related SAE, TEAE leading to death, TEAE leading to termination of trial, drug-relation TEAE leading to termination of trial and drug-related TEAE leading to discontinuation of use of test drug were summarized for case number, subject number and incidence rate. P value for the incidence of these AEs with different classifications was calculated by Fisher's exact test.

TEAE, SAE, drug-related TEAE, drug-related SAE, TEAE leading to the termination of the trial, and TEAE leading to the discontinuation of drug use were summarized and described according to the system organ classification (SOC), preferred terminology (PT) and study group. The severity of TEAE and drug-related TEAE was also summarized according to SOC, PT and study groups.

The measured value of parameters and changes from baseline of vital signs, 12-lead ECG, physical examination, clinical laboratory examination, etc. were summarized according to the planned time point and the study group.

Determine dose-limited toxicity of multiple dose in human (DLT); Determine the maximum tolerable dose of multiple dose in human (MTD).

ELIGIBILITY:
Subject inclusion criteria:

* Thalassemia patients with serum ferritin ≥ 500 µg/L
* Patients aged 16 and above
* HB≥80 g/L before administration
* Voluntarily participate in the experiment, and the process of obtaining informed consent met the requirements of GCP.

Subject exclusion criteria:

* Hepatitis B surface antigen positive, hepatitis B core antibody positive and HBV-DNA positive, hepatitis C anti-HCV positive, HIV positive, Treponema pallidum positive
* History of active digestive tract diseases (including gastric ulcer, duodenal ulcer, gastroesophageal varices, ulcerative colitis, Crohn's disease, digestive tract tumors, familial genetic polyps), history of digestive tract perforation, history of digestive tract surgery and influence on drug absorption, and other investigators believe that patients with potential intestinal complications
* Liver dysfunction (ALT or AST > 2.5×ULN); or renal dysfunction (serum creatinine > 1.5×ULN)
* Uncontrolled active infections
* Patients currently taking CYP3A strong inducer or inhibitor drugs or drugs that may prolong the QT interval without temporary suspension of use or temporary substitution of the said drugs
* Allergic constitution: allergic to or with contraindication of main ingredients or excipients of CN128 tablets (microcrystalline cellulose, cross-linked sodium carboxymethyl cellulose, silica, sodium stearate fumarate, Opadry)
* Patients who have abnormal ECG with clinical significance: congenital long QT syndrome or known family history of long QT syndrome; QTc > 450ms (male) or QTc > 470ms (female); patients who have ventricular or atrial tachyarrhythmia with clinical significance, etc
* Family planning participants (including male subjects) during or within three months after the trial
* Patients with a history of blood donation within 3 months before the trial
* Patients with a history of smoking (more than 5 cigarettes or products with equivalent nicotine per day), alcoholism (more than 14 units of alcohol per week: 1 alcohol unit equals 10 mL or 8 g pure alcohol; 25 mL 40% liquor, 330 mL 5% beer, 175 mL 12% red wine equals 1.0, 1.5, 2.0 alcohol units respectively), drug abuse and addiction history
* Patients who smoke, drink or eat any food containing alcohol, xanthine or grapefruit (including chocolate, tea, coffee or cola drinks) within 48 h before using of test drug
* The subjects should not join in other clinical drug or instrument study or some other clinical studies within 3 months before taking the study drug, except for non interventional studies;
* Patients with positive results of nicotine and urine drug screening
* Patients with difficulty in venous blood collection
* Patients with positive blood pregnancy test results
* Any patient with conditions which the investigators resume inappropriate to participate in this study, such as: poor health status, poor compliance, unwillingness or inability to comply with treatment regimens, including delayed visits

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Height (Unit: m) | Day 11
  The patient's height will be determined, and it's one kind of Physical examination.
Weight (Unit: kg) | Day 11
  The patient's weight will be determined, and it's one kind of Physical examination.
Generally Phisical examination | Day 11
  The patient's skin, neck, eyes, ears, nose, throat, chest, back, lymph nodes, arms, legs, nervous system, etc. will be observed, and it's one kind of Physical examination.
Pulse (Unit: bpm) | Day 1 to Day 11
  The patient's pulse will be determined, and it's one kind of vital signs checks.
Respiration (Unit: bpm) | Day 1 to Day 11
  The patient's respiration will be determined, and it's one kind of vital signs checks.
Blood pressure (Unit: mmHg) | Day 1 to Day 11
  Both patient's systolic and diastolic blood pressure will be measured, and it's one kind of vital signs checks.
Temperature (Unit: ℃) | Day 1 to Day 11
  The patient's temperature will be determined, and it's one kind of vital signs checks.
Electrocardiogram: P-R (Unit: ms), QRS (Unit: ms), QTc (Unit: ms), etc | Day 1 to Day 11
  The patient's electrocardiogram will be measured, and it's one kind of laboratory test.
WBC (Unit: 10E9/L), RBC (Unit: 10E9/L), NEUT (Unit: 10E9/L), BASO (Unit: 10E9/L) | Day 3, Day 7, Day 11
  The patient's blood examination（WBC (Unit: 10E9/L), RBC (Unit: 10E9/L), NEUT (Unit: 10E9/L), BASO (Unit: 10E9/L), etc.）will be determined at Day 3, Day 7, Day 11 respectively, and it's one kind of laboratory test.
ALT (Unit: U/L), AST (Unit: U/L) | Day 3, Day 7, Day 11
  The patient's blood biochemical examination（ALT (Unit: U/L), AST (Unit: U/L), etc.）will be determined at Day 3, Day 7, Day 11 respectively，and it's one kind of laboratory test.
Fibrinogen (Unit: g/L), Prothrombin time (Unit: s), APTT (Unit: s) | Day 11
  The patient's blood coagulation function ( fibrinogen (Unit: g/L), prothrombin time (Unit: s), APTT (Unit: s) , etc.) will be determined at Day 11, and it's one kind of laboratory test.
Serum iron (Unit: umol/L) | Day 11
  The patient's serum iron will be determined at Day 11, and it's one kind of laboratory test.
Urine colour | Day 3, Day 7, Day 11
  The colour of urine will be observed at Day 3, Day 7, Day 11 respectively，and it's one kind of laboratory test.
Urine appearance | Day 3, Day 7, Day 11
  The appearance of urine will be observed at Day 3, Day 7, Day 11 respectively，and it's one kind of laboratory test.
Urine glucose (Unit: mmol/L) | Day 3, Day 7, Day 11
  The glucose of urine will be determined at Day 3, Day 7, Day 11 respectively，and it's one kind of laboratory test.
Urine protein (Unit: g/L) | Day 3, Day 7, Day 11
  The protein of urine will be determined at Day 3, Day 7, Day 11 respectively，and it's one kind of laboratory test.
Number of subjects with adverse events | Day 1 to Day 11
  It's the number of subjects with adverse events after administration.
AUC0-t of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
AUC0-∞ of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Cmax of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Tmax of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
t1/2 of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
CL/F of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Vd/F of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
MRT of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Css-av of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Css-min of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Css-max of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Accumulation rate of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
Fluctuation index of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters
λz of CN128 | Day 1, Day 2, Day 3, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11
  Pharmacokinetics parameters

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China